CLINICAL TRIAL: NCT05568446
Title: Effectiveness of Social Virtual Reality Based Intervention on Enhancing Social Interaction Skills in Children With Attention-deficit/Hyperactivity Disorder: a Pilot Randomised Controlled Trial
Brief Title: Social VR Based Intervention on Enhancing Social Interaction Skills in Children With AD/HD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, WONG Portia, Principal Investigator, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HSEARS20220823001
Record Dates: First submitted 2022-09-30; First posted 2022-10-05 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
Keywords: Attention-deficit/hyperactivity disorder; Virtual reality; Social interaction skills; Children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Social VR group (Experimental): Social VR (SocVR) intervention is developed to enhance the social interaction skills of children. The participants will wear a head-mounted display (HMD) for the SocVR intervention. Each session of the SocVR intervention lasts for a maximum of 20 minutes to ensure the participants focus on the intervention and prevent causing any physical effect (Yamaguchi, 1999). The intervention contains three real-life virtual scenarios, including (1) classroom and playground, (2) MTR station and compartment, and (3) street and building. One scenario will be adopted in each session. The sequences of the scenarios used in each session will be the same for all participants. During the SocVR intervention, one RA will also appear as one avatar in the scenario to guide the participants to complete a series of tasks. Each intervention session will be conducted in a classroom independently for each participant.
  Interventions: Behavioral: Social virtual reality
- Traditional social skills group (Active Comparator): An experienced special educational needs (SEN) teacher will teach the participants social interaction skills through tradidactic instructions and role-play activities. Four modules will be covered in the 4-week training: (1) how to introduce yourself and basic social skills; (2) how to listen to others; (3) how to share with others; (4) learn to know how people feel and how to empathise. These modules have been applied in many studies (Braswell & Bloomquist, 1991; Huang et al., 2015). The content of this training will be as similar as possible to the SocVR training. The training lasts 20 minutes which depends on the emotion of the participants. Each training session will be conducted in a classroom independently for each participant.
  Interventions: Behavioral: Traditional social skills
- Waitlist control group (No Intervention): With reference to Beck et al. (2010), the participants in this group will receive no training and they can participate in the social VR training after the intervention period. To ensure the consistency of the experiment, the participants are not allowed to initiate or change their pharmacological treatment during the 8-week intervention period.

INTERVENTIONS:
Behavioral: Social virtual reality — The participants will receive eight training sessions in 4 weeks (2 sessions per week). Each session is about 20 minutes.
  Arms: Social VR group
Behavioral: Traditional social skills — The participants will receive eight training sessions in 4 weeks (2 sessions per week). Each session is about 20 minutes.
  Arms: Traditional social skills group

SUMMARY:
The study targets children with diagnosed ADHD and aims to (1) develop a social virtual reality based (SocVR) intervention and (2) investigate its effects on improving the social skills and executive functioning of inhibitions, emotional control and attention of the children compared to traditional social skills training.

The study will be a three-arm parallel randomised controlled trial comparing the effects of a SocVR with traditional social skills training on social skills and executive functioning of children with ADHD. The study period is 2 months, including 4 weeks (2 sessions per week) of intervention and control, followed by a 4-week follow-up. The participants will be assessed at three time points (i.e. at baseline, 4 weeks and 4 weeks follow-up).

The guidelines of Whitehead et al. (2016) suggested that recommended that at least 16 subjects per group for medium effect size in pilot RCT and 15% attrition over time can be expected. Thus, the minimum sample size per group was 20. A total of 60 participants will be recruited in which 20 participants in the social VR group, 20 in the traditional social skills group and 20 in the waitlist control group.

DETAILED DESCRIPTION:
Social VR Intervention During the Social VR intervention, one RA will also appear as one avatar in the scenario to guide the participants to complete a series of tasks. Each intervention session will be conducted in a classroom independently for each participant.

Traditional social skills training The training lasts 20 minutes which depends on the emotion of the participants. Each training session will be conducted in a classroom independently for each participant.

Sample size The guidelines of Whitehead et al. (2016) suggested that recommended that at least 16 subjects per group for medium effect size in pilot RCT and 15% attrition over time can be expected. Thus, the minimum sample size per group was 20. Based on the guideline of Whitehead et al. (2016), a total of 60 participants will be recruited in which 20 participants in the social VR group, 20 in the traditional social skills group and 20 in the waitlist control group. This sample size is comparable to those used in the published pilot study on children with ADHD. For instance, van der Oord et al. (2014) recruited 40 participants (20 in the control group and 20 in the interventional group) to examine the efficacy of computerized executive functioning remediation training with game elements in children with ADHD.

Recruitment Participants will be recruited from six primary schools and community centres. Interested participants or parents who provide written informed consent will be further evaluated for inclusion and exclusion criteria by a trained research assistant. Participants who meet the inclusion criteria in the study will be invited to perform an IQ test at the university at baseline.

Randomisation Eligible participants will be randomized to the SocVR group, traditional social skills training group or waitlist control group. A computer-generator randomiser will be used to generate the random allocation list. The randomisation will be undertaken by another research assistant not directly involved in the study. A number generated by the computer will be assigned to each eligible subject who will be randomly allocated to the three different groups by using the number. The participants and their parents or legal guardians will be blind to the assignment process. Parents or legal guardians will receive an email and a telephone call with notification to Group 1, Group 2 or Group 3.

Statistical analysis All statistical analyses will be performed in SPSS version 26.0 software (IBM Corp, Armonk, NY, USA) and are two-sided with a level of significance of < 0.05. Demographic information of the participants will be summarised with frequency and percentage for categorical variables. The continuous variables will be summarised by mean and standard deviation. The change between baseline and week 4 within each arm will be tested using t-tests. To examine the between-group difference in terms of measure outcomes from baseline to week 4, repeated analyses of covariance (ANCOVA) with adjustment of baseline characteristics will be conducted. To evaluate the improvement during the intervention period among the three groups, f-tests will be performed on primary and secondary outcome measures at the beginning of the first session and at the end of the last session. An intention-to-treat analysis will be performed. This analysis is regarded as the most appropriate approach to analyse RCT data by the highest-quality journals, which have utilised the CONSORT standard.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 6 and 12 years
* Ethnic Chinese
* Residing in Hong Kong
* Having received a diagnosis of ADHD by Child Assessment Service in Hong Kong or via private practice
* Stable on pharmacological and/or psychological treatment for ADHD 8 weeks before baseline (determined by health care professionals on the basis of medication data and behavioural observation)
* No initiation or change of pharmacological treatment for ADHD during the intervention period ability to read Chinese, and speak and listen to Cantonese by the child and by at least one of their parents or legal guardian
* Willing to provide informed consent by both participants and one of their parents or legal guardian

Exclusion Criteria:

* Comorbid autism
* Mental retardation
* An estimated IQ lower than 85 (using the Wechsler Intelligence Scale for Children - Fourth Edition (Hong Kong) (WISC-IV(HK)))
* Autism spectrum disorder (previously diagnosed by health care professionals)
* Comorbid acute psychiatric disorder (previously diagnosed by health care professionals)
* With a severe physical disability (e.g., blindness, deafness) or learning disability (e.g., dyslexia).

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-11-15 (Estimated); Primary Completion 2023-02-28 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Social Skills Rating Scale | Baseline
  This scale consists of 3 subscales, including self-control, assertiveness and initiative, and cooperation, with a total of 31 items. A 3-point Likert scale (never, sometimes, often) is used to score.
Social Skills Rating Scale | Change from baseline social skills at week 4 post-interventioin
  This scale consists of 3 subscales, including self-control, assertiveness and initiative, and cooperation, with a total of 31 items. A 3-point Likert scale (never, sometimes, often) is used to score.
Social Skills Rating Scale | Week 8 follow-up
  This scale consists of 3 subscales, including self-control, assertiveness and initiative, and cooperation, with a total of 31 items. A 3-point Likert scale (never, sometimes, often) is used to score.

SECONDARY OUTCOMES:
Behavior Rating Inventory of Executive Function | Baseline
  This scale is used to assess the executive functioning of children which will be scored by the participants' parents. The subscales of inhibitions (16-item), emotional control (10-item) and shifting (10-item) will be adopted in this study. A 3-point Likert scale (never, sometimes, often) is used to score.
Behavior Rating Inventory of Executive Function | Change from baseline social skills at week 4 post-interventioin
  This scale is used to assess the executive functioning of children which will be scored by the participants' parents. The subscales of inhibitions (16-item), emotional control (10-item) and shifting (10-item) will be adopted in this study. A 3-point Likert scale (never, sometimes, often) is used to score.
Behavior Rating Inventory of Executive Function | Week 8 follow-up
  This scale is used to assess the executive functioning of children which will be scored by the participants' parents. The subscales of inhibitions (16-item), emotional control (10-item) and shifting (10-item) will be adopted in this study. A 3-point Likert scale (never, sometimes, often) is used to score.

OTHER OUTCOMES:
Simulator Sickness Questionnaire | Week 4 post-interventioin
  This questionnaire measures the motion sickness or physical discomfort of the participants in the VR environment. Nine items will be measured, including general discomfort, fatigue, headache, eyestrain, sweating, nausea, difficulty concentrating, blurred vision and dizziness. Yes or no questions were used for each item.

CONTACTS AND LOCATIONS:
Overall Officials: Ka Po Wong, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The data will be available after the completion of the study writing.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).